CLINICAL TRIAL: NCT04429503
Title: A Randomized, Double-Masked, Active-Controlled Phase 2/3 Study of the Efficacy and Safety of High-Dose Aflibercept in Patients With Diabetic Macular Edema
Brief Title: Study of a High-Dose Aflibercept in Participants With Diabetic Eye Disease
Acronym: PHOTON
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGFTe-HD-DME-1934; 2019-003643-30 (EudraCT Number)
Record Dates: First submitted 2020-05-26; First posted 2020-06-12 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- aflibercept Q8 (Active Comparator): Administered every 8 weeks after a loading phase
  Interventions: Drug: aflibercept
- High-Dose aflibercept Q12 (Experimental): Administered every 12 weeks after a loading phase
  Interventions: Drug: High-dose aflibercept
- High-Dose aflibercept Q16 (Experimental): Administered every 16 weeks after a loading phase
  Interventions: Drug: High-dose aflibercept

INTERVENTIONS:
Drug: aflibercept — Intravitreally (IVT) administered as a liquid formulation in a vial
  Other Names: EYLEA®; BAY86-5321
  Arms: aflibercept Q8
Drug: High-dose aflibercept — Intravitreally (IVT) administered as a liquid formulation in a vial
  Arms: High-Dose aflibercept Q12; High-Dose aflibercept Q16

SUMMARY:
The primary objective of the study is to determine if treatment with high-dose aflibercept (HD) at intervals of 12 or 16 weeks provides non-inferior best corrected visual acuity (BCVA) compared to aflibercept dosed every 8 weeks.

The secondary objectives of the study are as follows:

* To determine the effect of HD vs. aflibercept on anatomic and other visual measures of response
* To evaluate the safety, immunogenicity, and pharmacokinetics (PK) of aflibercept

ELIGIBILITY:
Key Inclusion Criteria:

* Diabetic macular edema (DME) with central involvement in the study eye
* Best corrected visual acuity (BCVA) early treatment diabetic retinopathy study (ETDRS) letter score of 78 to 24 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye with decreased vision determined to be primarily the result of DME
* Willing and able to comply with clinic visits and study-related procedures
* Provide informed consent signed by study participant or legally acceptable representative

Extension Phase: All randomized patients that complete visit 26, week 96, as long as the patient 1) provides informed consent and 2) no treatment for DME has been given in the study eye other than the randomized study treatment.

Key Exclusion Criteria:

* Evidence of macular edema due to any cause other than diabetes mellitus in either eye
* Active proliferative diabetic retinopathy in the study eye
* IVT anti-VEGF treatment (aflibercept, ranibizumab, bevacizumab, brolucizumab, pegaptanib sodium) or panretinal laser photocoagulation (PRP) /macular laser photocoagulation within 12 weeks (84 days) or intraocular or periocular corticosteroids within 16 weeks (112 days) of the screening visit in the study eye
* Prior IVT investigational agents in either eye (eg, anti-ang-2/anti-VEGF bispecific monoclonal antibodies, gene therapy, etc.) at any time
* Treatment with ocriplasmin (JETREA®) in the study eye at any time

NOTE: Other Protocol Defined Inclusion/Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (129):
- United States (82):
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Arcadia, California
  - Regeneron Study Site, Beverly Hills, California
  - Regeneron Study Site, Campbell, California
  - Regeneron Study Site, Encino, California
  - Regeneron Study Site, Fullerton, California
  - Regeneron Study Site, Huntington Beach, California
  - Regeneron Study Site, Long Beach, California
  - Regeneron Study Site, Palo Alto, California
  - Regeneron Study Site, Pasadena, California
  - Regeneron Study Site, Poway, California
  - Regeneron Study Site, Rancho Cordova, California
  - Regeneron Study Site, Riverside, California
  - Regeneron Study Site, Torrance, California
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Durango, Colorado
  - Regeneron Study Site, Lakewood, Colorado
  - Regeneron Study Site, Waterford, Connecticut
  - Regeneron Study Site, Clearwater, Florida
  - Regeneron Study Site, Fort Lauderdale, Florida
  - Regeneron Study Site, Fort Myers, Florida
  - Regeneron Study Site, Jacksonville, Florida
  - Regeneron Study Site, Lakeland, Florida
  - Regeneron Study Site, Largo, Florida
  - Regeneron Study Site, Melbourne, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Pinellas Park, Florida
  - Regeneron Study Site, Plantation, Florida
  - Regeneron Study Site, St. Petersburg, Florida
  - Regeneron Study Site, Stuart, Florida
  - Regeneron Study Site, Winter Haven, Florida
  - Regeneron Study Site, Augusta, Georgia
  - Regeneron Study Site 1, Marietta, Georgia
  - Regeneron Study Site 2, Marietta, Georgia
  - Regeneron Study Site, ‘Aiea, Hawaii
  - Regeneron Study Site, Oak Forest, Illinois
  - Regeneron Study Site, Springfield, Illinois
  - Regeneron Study Site, Carmel, Indiana
  - Regeneron Study Site, Shawnee Mission, Kansas
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Hagerstown, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Royal Oak, Michigan
  - Regeneron Study Site, Southaven, Mississippi
  - Regeneron Study Site, Henderson, Nevada
  - Regeneron Study Site, Bloomfield, New Jersey
  - Regeneron Study Site, Edison, New Jersey
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, Great Neck, New York
  - Regeneron Study Site, Liverpool, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Oceanside, New York
  - Regeneron Study Site, Shirley, New York
  - Regeneron Study Site, Asheville, North Carolina
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Beachwood, Ohio
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Dublin, Ohio
  - Regeneron Study Site, Edmond, Oklahoma
  - Regeneron Study Site, Tulsa, Oklahoma
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Bethlehem, Pennsylvania
  - Regeneron Study Site, Kingston, Pennsylvania
  - Regeneron Study Site, Monroeville, Pennsylvania
  - Regeneron Study Site, Beaufort, South Carolina
  - Regeneron Study Site, Ladson, South Carolina
  - Regeneron Study Site, West Columbia, South Carolina
  - Regeneron Study Site, Rapid City, South Dakota
  - Regeneron Study Site, Germantown, Tennessee
  - Regeneron Study Site, Knoxville, Tennessee
  - Regeneron Study Site, Nashville, Tennessee
  - Regeneron Study Site, Abilene, Texas
  - Regeneron Study Site, Bellaire, Texas
  - Regeneron Study Site 2, San Antonio, Texas
  - Regeneron Study Site, The Woodlands, Texas
  - Regeneron Study Site, Willow Park, Texas
  - Regeneron Study Site 1, Salt Lake City, Utah
  - Regeneron Study Site, Fairfax, Virginia
  - Regeneron Study Site, Norfolk, Virginia
  - Regeneron Study Site, Morgantown, West Virginia
- Canada (4):
  - Regeneron Study Site, Calgary, Alberta
  - Regeneron Study Site, Mississauga, Ontario
  - Regeneron Study Site, North York, Ontario
  - Regeneron Study Site, Sherbrooke, Quebec
- Czechia (2):
  - Regeneron Study Site, Pardubice
  - Regeneron Study Site, Prague
- Germany (3):
  - Regeneron Study Site, Neubrandenburg, Mecklenburg-Westfalen
  - Regeneron Study Site, Göttingen, North Rhine-Westphalia
  - Regeneron Study Site, Münster, North Rhine-Westphalia
- Hungary (6):
  - Regeneron Study Site 1, Pécs, Baranya
  - Regeneron Study Site, Szombathely, Vas County
  - Regeneron Study Site, Zalaegerszeg, Zala County
  - Regeneron Study Site, Budapest
  - Regeneron Study Site, Debrecen
  - Regeneron Study Site, Szeged
- Japan (29):
  - Regeneron Study Site, Nagakute, Aichi-ken
  - Regeneron Study Site, Nagoya, Aichi-ken
  - Regeneron Study Site, Yoshida-Gun, Fukui
  - Regeneron Study Site, Kurume, Fukuoka
  - Regeneron Study Site, Kōriyama, Fukushima
  - Regeneron Study Site, Hakodate, Hokkaido
  - Regeneron Study Site, Kobe, Hyōgo
  - Regeneron Study Site, Mito, Ibaraki
  - Regeneron Study Site, Toride, Ibaraki
  - Regeneron Study Site, Tsuchiura-shi, Ibaraki
  - Regeneron Study Site, Kita-gun, Kagawa-ken
  - Regeneron Study Site, Kawasaki, Kanagawa
  - Regeneron Study Site, Matsumoto, Nagano
  - Regeneron Study Site, Nagasaki, Nagasaki
  - Regeneron Study Site, Kashihara, Nara
  - Regeneron Study Site, Hirakata, Osaka
  - Regeneron Study Site, Tokorozawa, Saitama
  - Regeneron Study Site, Susono, Shizuoka
  - Regeneron Study Site, Shimotsuke-shi, Tochigi
  - Regeneron Study Site, Chiyoda-ku, Tokyo
  - Regeneron Study Site, Hachiōji, Tokyo
  - Regeneron Study Site, Itabashi-ku, Tokyo
  - Regeneron Study Site, Meguro-ku, Tokyo
  - Regeneron Study Site, Ube, Yamaguchi
  - Regeneron Study Site, Fukuoka
  - Regeneron Study Site, Kagoshima
  - Regeneron Study Site, Osaka
  - Regeneron Study Site, Saitama
  - Regeneron Study Site, Tokushima
- Regeneron Study Site, Arecibo, Puerto Rico
- United Kingdom (2):
  - Regeneron Study Site, Sunderland, Tyne and Wear
  - Regeneron Study Site, London

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to study documents (including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan) that support the methods and findings reported in a manuscript. Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification.
URL: https://vivli.org/

REFERENCES:
- [Derived] Suzuma K, Murata T, Shimura M, Yoshida S, Kishino G, Berliner AJ, Chu KW, Reed K, Vitti R, Cheng Y, Voronca D, Bhore R, Leal S, Morgan-Warren P, Schulze A, Schmidt-Ott U, Kobayashi M, Sakamoto T; PHOTON Investigators. Intravitreal aflibercept 8 mg in patients from Japan with diabetic macular edema: 48-week subgroup analysis of the PHOTON trial. Jpn J Ophthalmol. 2025 Dec 26. doi: 10.1007/s10384-025-01271-7. Online ahead of print. PMID 41452566
- [Derived] Do DV, Wykoff CC, Sivaprasad S, Brown DM, Boyer DS, Sakamoto T, Win P, Joshi S, Salehi-Had H, Seres A, Berliner AJ, Leal S, Vitti R, Chu KW, Reed K, Cheng Y, Bhore R, Bai Z, Schmidt-Ott U, Schmelter T, Schulze A, Hasanbasic Z, Morgan-Warren PJ, Zhang X, Hirshberg B, Yancopoulos GD; PHOTON Investigators. Intravitreal Aflibercept 8 mg for Diabetic Macular Edema: Ninety-Six-Week Results from the Randomized Phase 2/3 PHOTON Trial. Ophthalmology. 2025 Nov 10:S0161-6420(25)00707-9. doi: 10.1016/j.ophtha.2025.10.028. Online ahead of print. PMID 41223900
- [Derived] Brown DM, Boyer DS, Do DV, Wykoff CC, Sakamoto T, Win P, Joshi S, Salehi-Had H, Seres A, Berliner AJ, Leal S, Vitti R, Chu KW, Reed K, Rao R, Cheng Y, Sun W, Voronca D, Bhore R, Schmidt-Ott U, Schmelter T, Schulze A, Zhang X, Hirshberg B, Yancopoulos GD, Sivaprasad S; PHOTON Investigators. Intravitreal aflibercept 8 mg in diabetic macular oedema (PHOTON): 48-week results from a randomised, double-masked, non-inferiority, phase 2/3 trial. Lancet. 2024 Mar 23;403(10432):1153-1163. doi: 10.1016/S0140-6736(23)02577-1. Epub 2024 Mar 7. PMID 38461843

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 970 participants were screened and 660 participants were randomized, of whom 658 participants received at least 1 dose of study treatment in the study eye. Fellow eye treatment was allowed with 2 mg aflibercept at the investigator's discretion for indications approved by governing authorities. The treated fellow eye was not considered an additional study eye. Only one study eye per participant was analyzed within the study.
Groups:
- Aflibercept 2 mg Every 8 Weeks (2q8): Participants received 2 milligrams (mg) aflibercept every 8 weeks (2q8), following 5 initial monthly doses
- High-dose (HD) Aflibercept Every 12 Weeks (HDq12): Participants received HD aflibercept (8 mg) every 12 weeks (HDq12) following 3 initial monthly doses
- HD Aflibercept Every 16 Weeks (HDq16): Participants received HD aflibercept (8mg) every 16 weeks (HDq16) following 3 initial monthly doses
- 2q8/HD Aflibercept (Extension): Participants receiving aflibercept 2q8 switched to HD in the extension phase
- HDq12 Aflibercept (Extension): Participants continued to receive HDq12 aflibercept during the extension phase
- HDq16 Aflibercept (Extension): Participants continued to receive HDq16 aflibercept during the extension phase
Period: Main Study (Up to Wk 96)
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16) | 2q8/HD Aflibercept (Extension) | HDq12 Aflibercept (Extension) | HDq16 Aflibercept (Extension)
Started (Randomized) | 167 | 329 | 164 | 0 | 0 | 0
Treated (All randomized participants who received at least 1 dose of study drug (Full Analysis Set)) | 167 | 328 | 163 | 0 | 0 | 0
Completed Week 48 | 157 | 300 | 156 | 0 | 0 | 0
Completed Week 60 | 155 | 289 | 152 | 0 | 0 | 0
Completed (Completed Week 96) | 139 | 256 | 139 | 0 | 0 | 0
Not Completed | 28 | 73 | 25 | 0 | 0 | 0
Not completed — Non-compliance with protocol by the subject | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 9 | 2 | 0 | 0 | 0
Not completed — Decision by the investigator/sponsor | 2 | 9 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 17 | 8 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 19 | 7 | 0 | 0 | 0
Not completed — Death | 9 | 18 | 5 | 0 | 0 | 0
Period: Extension Phase (Wk 96 to Wk 156)
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16) | 2q8/HD Aflibercept (Extension) | HDq12 Aflibercept (Extension) | HDq16 Aflibercept (Extension)
Started (Number of participants treated during extension phase) | 0 | 0 | 0 | 70 | 130 | 65
Completed (Number of participants who completed Week 156 (End of Study)) | 0 | 0 | 0 | 58 | 103 | 49
Not Completed | 0 | 0 | 0 | 12 | 27 | 16
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Decision by the Investigator/Sponsor | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 10 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 6 | 6
Not completed — Death | 0 | 0 | 0 | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug; it was based on the treatment assigned to the participant at baseline (as randomized). Only one study eye per participant was analyzed within the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16) | Total
Number analyzed (Participants) | 167 | 328 | 163 | 658
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.78) | 62.1 (11.13) | 61.9 (9.50) | 62.3 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 118 | 64 | 257
  Male | 92 | 210 | 99 | 401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 54 | 34 | 119
  Not Hispanic or Latino | 133 | 266 | 126 | 525
  Unknown or Not Reported | 3 | 8 | 3 | 14
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 2 | 0 | 2
    Asian | 30 | 48 | 23 | 101
    Black or African American | 18 | 35 | 9 | 62
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    White | 112 | 231 | 128 | 471
    Multiple | 0 | 1 | 0 | 1
    Other | 4 | 6 | 1 | 11
    Not Reported | 3 | 4 | 2 | 9
Best Corrected Visual Acuity (BCVA) in the Study Eye [Mean (Standard Deviation); unit: Letters] — Early Treatment Diabetic Retinopathy Study (ETDRS) letter score; Only one study eye per participant was analyzed within the study
  Letters | 61.5 (11.22) | 63.6 (10.10) | 61.4 (11.76) | 62.5 (10.86)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) (Early Treatment Diabetic Retinopathy Study [ETDRS] Letter Score) in the Study Eye at Week 48
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. BCVA scale range is 0 (worst) to 100 (best).
Time Frame: Baseline, Week 48
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug; it was based on the treatment assigned to the participant at baseline (as randomized); Only one study eye per participant was analyzed within the study.
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
Letters | 8.67 (0.73) | 8.10 (0.61) | 7.23 (0.71)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Every 8 Weeks (2q8) vs High-dose (HD) Aflibercept Every 12 Weeks (HDq12); Test type: Non-Inferiority — p-value for one-sided non-inferiority (NI) test at a margin of 4 letters; p < 0.0001, Mixed Model for Repeated Measurements; Least Square (LS) Mean Difference = -0.57, 95% CI 2-sided [-2.26 to 1.13] — HDq12 minus 2q8
Statistical Analysis 2: Comparison: Aflibercept 2 mg Every 8 Weeks (2q8) vs HD Aflibercept Every 16 Weeks (HDq16); Test type: Non-Inferiority — p-value for one-sided non-inferiority (NI) test at a margin of 4 letters; p = 0.0031, Mixed Model for Repeated Measurements; LS Mean Difference = -1.44, 95% CI 2-sided [-3.27 to 0.39] — HDq16 minus 2q8

2. Secondary Outcome: Percentage of Participants With a ≥2 Step Improvement From Baseline in Diabetic Retinopathy Severity Scale (DRSS) Score at Week 48
Description: The DRSS was assessed according to the following scale: 10 = Diabetic retinopathy (DR) absent, 14 = DR questionable, 15 = DR questionable, 20 = Micro-aneurysms only, 35 = Mild Non-proliferative diabetic retinopathy (NPDR), 43 = Moderate NPDR, 47 = Moderately severe NPDR, 53 = Severe NPDR, 61 = Mild Proliferative diabetic retinopathy (PDR), 65 = Moderate PDR, 71 = High-risk PDR, 75 = High-risk PDR, 81 = Advanced PDR: fundus partially obscured, center of macula attached, 85 = Advanced PDR: posterior fundus obscured, or center of macula detached, 90 = cannot grade, even sufficiently for level 81 or 85.
Time Frame: Baseline, Week 48
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug; it was based on the treatment assigned to the participant at baseline (as randomized); Only one study eye per participant was analyzed within the study,
Measure: Number; unit: Percentage of Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 158 | 310 | 153
Percentage of Participants | 26.6 | 29.0 | 19.6
Statistical Analysis 1: Comparison: Aflibercept 2 mg Every 8 Weeks (2q8) vs High-dose (HD) Aflibercept Every 12 Weeks (HDq12); Test type: Non-Inferiority — The non-inferiority margin was set at 15%; Adjusted Difference (%) = 1.98, 95% CI 2-sided [-6.61 to 10.57] — Difference with confidence interval (CI) was calculated using Mantel-Haenszel weighting scheme adjusted for stratification factors
Statistical Analysis 2: Comparison: Aflibercept 2 mg Every 8 Weeks (2q8) vs HD Aflibercept Every 16 Weeks (HDq16); Test type: Non-Inferiority — The non-inferiority margin was set at 15%; Adjusted Difference (%) = -7.52, 95% CI 2-sided [-16.88 to 1.84] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline at Week 48
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. BCVA scale range is 0 (worst) to 100 (best). Only one study eye per participant was analyzed within the study
Time Frame: Baseline, Week 48
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug; it was based on the treatment assigned to the participant at baseline (as randomized)
Measure: Number; unit: Percentage of Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 165 | 326 | 163
Percentage of Participants | 23.0 | 18.7 | 16.6

4. Secondary Outcome: Percentage of Participants With BCVA ≥69 Letters at Week 48
Description: as for outcome 1
Time Frame: At Week 48
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 165 | 326 | 163
Percentage of Participants | 63.0 | 65.3 | 62.6

5. Secondary Outcome: Percentage of Participants Without Fluid at Foveal Center at Week 48
Description: Retinal fluid status was evaluated using spectral domain optical coherence tomography (SD-OCT) on the study eye.
Time Frame: At Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 165 | 325 | 162
Percentage of Participants | 54.5 | 58.5 | 43.8

6. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye at Week 48
Description: Central Retinal Thickness (CRT) was measured in the study eye by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Baseline, Week 48
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Microns
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
Microns | -164.85 (8.79) | -176.77 (5.73) | -148.84 (9.45)

7. Secondary Outcome: Percentage of Participants Without Leakage on Fluorescein Angiography (FA) at Week 48
Description: Leakage is the release of fluorescein dye from diseased retinal vessels.
Time Frame: At Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 162 | 303 | 152
Percentage of Participants | 2.5 | 7.6 | 0.7

8. Secondary Outcome: Change From Baseline in National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) Total Score at Week 48
Description: Vision-specific quality of life is assessed with the NEI VFQ-25 (National Eye Institute Visual Function Questionnaire), i.e. a 25-item questionnaire that gives a score on a scale from 0 (worst) to 100 (best = no vision problems).
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
Score on a Scale | 2.82 (1.10) | 4.06 (0.80) | 2.94 (0.93)

9. Secondary Outcome: Systemic Pharmacokinetics (PK) of Aflibercept as Assessed by Plasma Concentrations Through Week 48
Description: Concentrations of Free Aflibercept in Plasma by Time and Treatment Group
Time Frame: Through Week 48
Population: Pharmacokinetic analysis set (PKAS): All treated participants who received any amount of study drug and had at least 1 non-missing free or bound aflibercept measurement following the first dose of study drug as applicable. The PKAS is based on the actual treatment received (as treated) rather than as randomized.
Measure: Mean (Standard Deviation); unit: milligram/Litre (mg/L)
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
milligram/Litre (mg/L) | 0.00102 (0.00580) | 0.0111 (0.0157) | 0.00105 (0.00477)

10. Secondary Outcome: Change From Baseline in BCVA in the Study Eye in Participants With Both Baseline and Week 48 BCVA
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. BCVA scale range is 0 (worst) to 100 (best). (Per Statistical Analysis Plan (SAP) Version 2.0 Appendix 10.9 for US Only)
Time Frame: Baseline, Week 48
Population: Full Analysis Set (FAS) - for participants who had both baseline BCVA and week 48 BCVA; Only one study eye per participant was analyzed within the study
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 153 | 291 | 154
Letters | 9.11 (8.94) | 9.14 (8.35) | 9.11 (7.30)

11. Secondary Outcome: Change From 8-weeks Post Initial Treatment Phase in BCVA in the Study Eye in Participants With Both 8-weeks Post Initial Treatment Phase BCVA and Week 48 BCVA
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. BCVA scale range is 0 (worst) to 100 (best). (Per SAP Version 2.0 Appendix 10.9 for US Only)
Time Frame: Baseline, Week 48
Population: Full Analysis Set (FAS) - for participants who had both BCVA at 8 weeks post initial treatment and week 48 BCVA; Only one study eye per participant was analyzed within the study
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 152 | 282 | 153
Letters | 1.63 (6.65) | 1.68 (5.54) | 1.64 (4.75)

12. Secondary Outcome: Change From Baseline in BCVA (Region-specific Analysis) in the Study Eye at Week 60
Description: as for outcome 1
Time Frame: Baseline, Week 60
Population: FAS: All randomized participants who received at least 1 dose of study drug; it was based on the treatment assigned to the participant at baseline (as randomized); Here, Number of Participants Analyzed = Number of participants with week 60 data. Only one study eye per participant was analyzed within the study
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
Letters | 9.40 (0.77) | 8.52 (0.63) | 7.64 (0.75)

13. Secondary Outcome: Assessment of Immunogenicity to Aflibercept by Measuring the Incidence of Treatment-emergent Anti-drug Antibodies (ADA) Response Through Week 96
Description: Number of participants with pre-existing immunoreactivity and treatment-emergent ADA response reported
Time Frame: Through Week 96
Population: ADA analysis set (AAS): All treated participants who received any amount of study drug and had at least 1 non-missing anti-aflibercept antibody result following the first dose of study drug. The AAS is based on the actual treatment received (as treated) rather than as randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 151 | 289 | 150
Participants
  Pre-existing Immunoreactivity | 4 | 11 | 2
  Treatment-Emergent | 2 | 7 | 4

14. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) Through Week 96
Description: A TEAE is an AE starting after the first dose of study drug to the last dose of study drug (active or sham) plus 30 days. Additionally, for patients who are still participating in the study (ie, have not been withdrawn and are continuing in the extension phase of the study) as of the week 96 visit all AEs up through the date of the week 96 visit were considered treatment-emergent.
Time Frame: Through Week 96
Population: Safety analysis set (SAF): All randomized participants who received any study treatment; it was based on the treatment received (as treated)
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
Participants | 134 | 277 | 143

15. Secondary Outcome: Number of Participants With Any Serious TEAE Through Week 96
Description: as for outcome 14
Time Frame: Through Week 96
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | High-dose (HD) Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16)
Number analyzed (Participants) | 167 | 328 | 163
Participants | 46 | 81 | 44

16. Secondary Outcome: Number of Participants With Any TEAE Through Week 156
Description: TEAEs are defined as AEs starting after the first dose of study drug to the last dose of study drug (active or sham) plus 30 days or week 156 visit, whichever was later.
Time Frame: Through Week 156
Population: Extension Safety Analysis Set (eSAF): All participants in the SAF who enrolled in the extension phase and completed the extension baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 2q8/HD Aflibercept (Extension) | HDq12 Aflibercept (Extension) | HDq16 Aflibercept (Extension)
Number analyzed (Participants) | 70 | 130 | 65
Participants | 64 | 122 | 59

17. Secondary Outcome: Number of Participants With Any Serious TEAE Through Week 156
Time Frame: Through Week 156
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | 2q8/HD Aflibercept (Extension) | HDq12 Aflibercept (Extension) | HDq16 Aflibercept (Extension)
Number analyzed (Participants) | 70 | 130 | 65
Participants | 27 | 41 | 22

ADVERSE EVENTS:
Time Frame: From first study treatment through week 156
Groups:
- Aflibercept 2 mg Every 8 Weeks (2q8); HD Aflibercept Every 12 Weeks (HDq12); HD Aflibercept Every 16 Weeks (HDq16): (baseline through week 96)
- 2q8/HD Aflibercept (Extension): Participants receiving aflibercept 2q8 switched to HD in the extension phase (week 96 through week 156)
- HDq12 Aflibercept (Extension): Participants continued to receive HDq12 aflibercept during the extension phase (week 96 through 156)
- HDq16 Aflibercept (Extension): Participants continued to receive HDq16 aflibercept during the extension phase (week 96 through 156)
Arm/Group | Aflibercept 2 mg Every 8 Weeks (2q8) | HD Aflibercept Every 12 Weeks (HDq12) | HD Aflibercept Every 16 Weeks (HDq16) | 2q8/HD Aflibercept (Extension) | HDq12 Aflibercept (Extension) | HDq16 Aflibercept (Extension)
All-Cause Mortality (participants affected / at risk) | 9/167 | 18/328 | 5/163 | 2/70 | 7/130 | 3/65
Serious Adverse Events (participants affected / at risk) | 46/167 | 84/328 | 45/163 | 27/70 | 46/130 | 23/65
Other Adverse Events (participants affected / at risk) | 98/167 | 190/328 | 116/163 | 50/70 | 99/130 | 50/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Every 8 Weeks (2q8) (N=167) | HD Aflibercept Every 12 Weeks (HDq12) (N=328) | HD Aflibercept Every 16 Weeks (HDq16) (N=163) | 2q8/HD Aflibercept (Extension) (N=70) | HDq12 Aflibercept (Extension) (N=130) | HDq16 Aflibercept (Extension) (N=65)
COVID-19 (Infections and infestations) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (4) | 5 (5) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 10 (10) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 7 (7) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract Fellow Eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diabetic retinopathy Fellow Eye (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Retinal haemorrhage Fellow Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage Fellow Eye (Eye disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (3) | 1 (3) | 0 (0)
Retinal artery occlusion Fellow Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tractional retinal detachment Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract subcapsular Study Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment Study Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis Study Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage Study Eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased Study Eye (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiretinal membrane Fellow Eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased Fellow Eye (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear Study Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract Study Eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Retinal neovascularisation Study Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis Study Eye (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear Study Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Occipital lobe stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Every 8 Weeks (2q8) (N=167) | HD Aflibercept Every 12 Weeks (HDq12) (N=328) | HD Aflibercept Every 16 Weeks (HDq16) (N=163) | 2q8/HD Aflibercept (Extension) (N=70) | HDq12 Aflibercept (Extension) (N=130) | HDq16 Aflibercept (Extension) (N=65)
COVID-19 (Infections and infestations) | 15 (16) | 40 (41) | 26 (27) | 6 (6) | 19 (22) | 15 (18)
Hypertension (Vascular disorders) | 22 (31) | 35 (38) | 31 (34) | 6 (10) | 21 (22) | 13 (13)
Cataract Fellow Eye (Eye disorders) | 8 (8) | 17 (17) | 14 (14) | 7 (7) | 18 (19) | 8 (8)
Cataract Study Eye (Eye disorders) | 5 (5) | 18 (19) | 18 (18) | 8 (8) | 18 (18) | 10 (10)
Vitreous floaters Study Eye (Eye disorders) | 6 (6) | 19 (20) | 7 (8) | 3 (3) | 8 (9) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 12 (12) | 9 (9) | 2 (2) | 5 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6) | 9 (12) | 2 (2) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (11) | 21 (24) | 10 (12) | 5 (7) | 16 (21) | 4 (7)
Urinary tract infection (Infections and infestations) | 10 (12) | 9 (13) | 7 (8) | 4 (6) | 8 (10) | 1 (1)
Conjunctival haemorrhage Study Eye (Eye disorders) | 6 (7) | 18 (18) | 8 (9) | 2 (3) | 4 (5) | 3 (4)
Coronary artery disease (Cardiac disorders) | 4 (4) | 5 (5) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Eye pain Study Eye (Eye disorders) | 4 (4) | 10 (10) | 3 (3) | 2 (2) | 3 (3) | 4 (5)
Punctate keratitis Study Eye (Eye disorders) | 1 (1) | 5 (5) | 7 (7) | 1 (1) | 3 (3) | 5 (5)
Retinal haemorrhage Study Eye (Eye disorders) | 1 (1) | 0 (0) | 6 (7) | 1 (1) | 1 (1) | 5 (6)
Vision blurred Study Eye (Eye disorders) | 5 (5) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Visual acuity reduced Study Eye (Eye disorders) | 4 (4) | 6 (9) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Visual impairment Study Eye (Eye disorders) | 1 (1) | 6 (6) | 3 (3) | 0 (0) | 4 (4) | 4 (4)
Vitreous detachment Study Eye (Eye disorders) | 7 (7) | 16 (16) | 5 (5) | 3 (3) | 8 (8) | 2 (2)
Intraocular pressure increased Study Eye (Eye disorders) | 7 (13) | 9 (12) | 2 (2) | 5 (15) | 2 (2) | 2 (2)
Diabetic retinal oedema Fellow Eye (Eye disorders) | 6 (7) | 15 (17) | 8 (8) | 5 (6) | 8 (8) | 3 (3)
Punctate keratitis Fellow Eye (Eye disorders) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 4 (5)
Vitreous detachment Fellow Eye (Eye disorders) | 7 (7) | 7 (8) | 5 (5) | 3 (3) | 4 (4) | 4 (4)
Vitreous floaters Fellow Eye (Eye disorders) | 4 (4) | 4 (4) | 8 (9) | 2 (2) | 3 (3) | 5 (7)
Vitreous haemorrhage Fellow Eye (Eye disorders) | 5 (5) | 7 (10) | 6 (7) | 6 (10) | 8 (11) | 3 (4)
Diabetic retinopathy Fellow Eye (Eye disorders) | 5 (5) | 5 (6) | 9 (9) | 2 (2) | 3 (3) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 8 (8) | 6 (6) | 0 (0) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 5 (7) | 5 (6) | 6 (6) | 4 (5) | 2 (3) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 5 (5) | 3 (3) | 5 (6) | 5 (5) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 8 (8) | 3 (3) | 0 (0) | 3 (3) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 2 (3) | 2 (3) | 5 (5) | 1 (1) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (7) | 8 (8) | 8 (8) | 4 (5) | 3 (3) | 5 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 10 (10) | 7 (7) | 0 (0) | 5 (5) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (9) | 5 (5) | 3 (3) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 11 (12) | 5 (5) | 4 (5) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 13 (16) | 4 (4) | 3 (4) | 8 (8) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 6 (6) | 2 (2) | 4 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT04429503/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT04429503/SAP_001.pdf